CLINICAL TRIAL: NCT04968483
Title: A Prospective Study of Perioperative Nutritional Status and Nutritional Support in Patients With Spinal Deformity
Brief Title: Perioperative Nutritional Status and Nutritional Support in Patients With Spinal Deformity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2020093
Record Dates: First submitted 2021-07-01; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Spine Deformity
Keywords: Spine deformity, Nutritional support, Postoperative complications
MeSH Terms: conditions — Postoperative Complications | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients with spine deformity undergoing surgical treatment
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — The general data, data of postoperative complications, data of nutritional assessment and nutritional support will be collected.

SUMMARY:
To investigate the nutritional status, nutritional support and postoperative complications of patients undergoing spinal orthopedic surgery during the perioperative period.

DETAILED DESCRIPTION:
Adopting the method of continuous fixed point sampling, the inpatients in the orthopedic ward of our hospital were selected as the objects of investigation.

(1) Data collection

1. general data: The information of gender, age, ethnicity, height, weight, course of disease, family history, combined diseases, medication etc.
2. Nutritional assessment：①Nutritional risk screening tool 2002(NRS 2002), an evidence-based nutritional risk screening tool developed by the European Society for Parenteral and Endoenteral Nutrition, was recommended by the Chinese Society for Parenteral and Endoenteral Nutrition as a nutritional risk screening tool for inpatients in China. The total NRS 2002 was divided into three scores, namely disease severity score, impaired nutritional status score and age score. NRS 2002 score ≥3 (accompanied by poor general conditions, such as weight loss, appetite, mental state, etc.) are at nutritional risk and require nutritional support; Those with a score less than 3 have no nutritional risk and do not need nutritional support. ②Other indicators include height, weight and body mass index, as well as biochemical indicators such as pre-albumin and hemoglobin. Nutritional assessment was performed within 24 hours of admission, on the 1d after surgery, on the 7d after surgery, every 7d after surgery, or upon discharge. NRS 2002 was repeated to assess patients' nutritional risk at the first review three months after discharge.
3. Nutritional support: The nutritional support received during the hospital was recorded, including the form of nutritional support (enteral or parenteral nutrition), energy ratio, variety selection, duration of administration, etc. 1 g carbohydrate provided 16.74 kJ(4 kcal) calories, 1 g fat milk provided 38.93 kJ(9.3 kcal) calories and 1 g amino acid provided 16.74 kJ(4 kcal) calories to calculate the energy provided by the nutritional support program. The amount of nitrogen provided by the nutritional support program was calculated with about 1 g nitrogen provided by 6.25 g amino acids.
4. Complications: Postoperative complications, such as sepsis, pneumonia, urinary tract infection, wound infection, and delayed wound healing, were recorded during hospitalization and within 3 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spine deformity, complete the operation in one time；
* Age: More than 10 years old ；
* Patients and their family members agreed to participate in the study and signed the informed consent；
* Conscious, patient or family members can communicate verbally.

Exclusion Criteria:

* Emergency surgery；
* Hospital stay less than 24 hours；
* Surgery was not performed during the hospital stay；
* Nutritional metabolic diseases.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Orthopaedic patients with spine deformity
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Data of nutritional assessment and support | Through the hospitalization, an average of 10 days.
  NRS2002 nutritional assessment results
Blood parameters about nutritional assessment and support | Baseline
  Hemoglobin values
Blood parameters about nutritional assessment and support | Through the hospitalization after surgery, an average of 10 days.
  blood hemoglobin values
Blood parameters about nutritional assessment and support | Baseline
  blood prealbumin values
Blood parameters about nutritional assessment and support | Through the hospitalization after surgery, an average of 10 days.
  Prealbumin values

SECONDARY OUTCOMES:
Complication rate | After surgery to 3-month follow-up
  Postoperative complication rate during hospitalization and within 3 months after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Ruifeng Xu, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No